CLINICAL TRIAL: NCT00076336
Title: Randomized, Double-Blind Trial of Telbivudine Versus Lamivudine in Adults With Decompensated Chronic Hepatitis B and Evidence of Cirrhosis
Brief Title: Telbivudine Versus Lamivudine in Adults With Decompensated Chronic Hepatitis B and Evidence of Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLDT600A2301
Record Dates: First submitted 2004-01-20; First posted 2004-01-22 (Estimated); Results first posted 2011-09-05 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-08

CONDITIONS: Hepatitis; Hepatitis B, Chronic; Cirrhosis
MeSH Terms: conditions — Hepatitis; Hepatitis B, Chronic; Fibrosis | interventions — Telbivudine; Lamivudine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Telbivudine 600 mg (Experimental): Participants received Telbivudine 600 mg and a matching lamivudine placebo orally once a day for up to 104 weeks. Participants were followed-up for 16 weeks post-treatment.
  Interventions: Drug: Telbivudine; Drug: Placebo
- Lamivudine 100 mg (Active Comparator): Lamivudine 100 mg and a Telbivudine matching placebo orally once a day for up to 104 weeks. Participants were followed-up for 16 weeks post-treatment.
  Interventions: Drug: Lamivudine; Drug: Placebo

INTERVENTIONS:
Drug: Telbivudine — 600mg/day oral tablet for 104 weeks
  Other Names: LDT600
  Arms: Telbivudine 600 mg
Drug: Lamivudine — 100mg/day oral tablet for 104 weeks
  Arms: Lamivudine 100 mg
Drug: Placebo — Telbivudine matching placebo or lamivudine matching placebo tablet.

SUMMARY:
This research study was conducted to compare the safety and effectiveness of the investigational medication, LdT (Telbivudine) versus Lamivudine, a drug currently approved by the US, European and Asian Health Authorities for the treatment of Hepatitis B infection. The results for patients taking LdT will be compared to results for patients taking lamivudine.

DETAILED DESCRIPTION:
Multicenter, multinational, randomized, double-blind study designed to compare the safety and efficacy of telbivudine (600 mg/day) versus lamivudine (100 mg/day) for 104 weeks in adults with decompensated chronic hepatitis B and evidence of cirrhosis. Patients were pre-stratified by screening Child-Turcotte-Pugh score (CTP score < 9 or ≥ 9) and ALT level (within normal limits (WNL) or > 1.0 x ULN) to help assure similar degrees of hepatic insufficiency and liver inflammation on both treatment arms. After 104 weeks of treatment, participants were followed-up with for an additional 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Documented decompensated chronic hepatitis B defined by all of the following: 1. Clinical history compatible with decompensated chronic hepatitis B related cirrhosis; 2. Child-Turcotte-Pugh score > 7 points.
* Evidence of hepatic cirrhosis or portal hypertension.

Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Patient is pregnant or breastfeeding.
* Patient is coinfected with hepatitis C virus (HCV), hepatitis D virus (HDV), or Human immunodeficiency virus (HIV).
* Patient previously received lamivudine, adefovir, or an investigational anti-hepatitis B virus (HBV) nucleoside or nucleotide analog at any time
* Patient has received interferon or other immunomodulatory treatment for HBV infection in the 12 months before Screening for this study.

Other protocol-defined exclusion criteria may apply.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2003-12; Primary Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (8):
  - Phoenix, Arizona
  - Los Angeles, California
  - Denver, Colorado
  - Indianapolis, Indiana
  - Rochester, Minnesota
  - New York, New York
  - Houston, Texas
  - Madison, Wisconsin
- Heidelburg, Australia
- Winnipeg, Canada
- Hong Kong, China
- Villejuif, France
- Hanover, Germany
- Novartis, New Delhi, India
- Tel Aviv, Israel
- Novartis, Riga, Latvia
- Novartis, Kuala Lumpur, Malaysia
- Auckland, New Zealand
- Novartis, Krakow, Poland
- Novartis, Moscow, Russia
- Singapore, Singapore
- Seoul, South Korea
- Barcelona, Spain
- Taipei, Taiwan
- Bangkok, Thailand
- Novartis, Istanbul, Istanbul, Turkey (Türkiye)
- London, United Kingdom
- Novartis, Hanoi, Vietnam

REFERENCES:
- [Result] E.J. Gane, H.L. Chan, G. Choudhuri, D.J. Suh4, A. Chutaputti, R. Safadi, T. Tanwandee, S. Thongsawat, N. Assy, S.K. Sarin, W. Bao, A. Trylesinski, C. Avila. TREATMENT OF DECOMPENSATED HBV-CIRRHOSIS: RESULTS FROM 2-YEARS RANDOMIZED TRIAL WITH TELBIVUDINE OR LAMIVUDINE. Journal of Hepatology 52, Supplement 1, Page S4. April 2010

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 232 patients randomized. One randomized patient in the telbivudine treatment group discontinued prior to commencing treatment and was excluded from the intent to treat (ITT) population. Three randomized patients (two in lamivudine group and one in telbivudine group) had no HBV DNA assessments after baseline and were excluded from ITT population.
Groups:
- Telbivudine 600 mg: Participants received Telbivudine 600 mg and a matching placebo to lamivudine orally once a day for up to 104 weeks, followed by a 16-week follow-up period.
- Lamivudine 100 mg: Participants received Lamivudine 100 mg and matching placebo to Telbivudine orally once a day for up to 104 weeks, followed by a 16-week follow-up period.
Period: Overall Study
Arm/Group | Telbivudine 600 mg | Lamivudine 100 mg
Started | 116 | 116
Safety Population | 115 (1 patient was randomized but never received study drug and not included in safety population.) | 116
Intent to Treat (ITT) Population | 114 (1 patient had no HBV DNA assessments after baseline and was excluded from ITT population.) | 114 (2 patients had no HBV DNA assessments after baseline and were excluded from ITT population.)
Completed Week 52 | 97 | 94
Completed Week 104 | 70 | 62
Completed | 64 | 60
Not Completed | 52 | 56
Not completed — Death | 13 | 17
Not completed — Adverse Event | 4 | 4
Not completed — Lost to Follow-up | 4 | 4
Not completed — Non-Compliance | 2 | 0
Not completed — Creatinine Clearance < 30 or Dialysis | 0 | 1
Not completed — Patient, Investigator, Sponsor request | 8 | 6
Not completed — Liver Transplantation | 3 | 3
Not completed — Virologic Breakthrough | 14 | 16
Not completed — Treatment failure | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telbivudine 600 mg | Lamivudine 100 mg | Total
Number analyzed (Participants) | 114 | 114 | 228
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline measures are based on intention to treat (ITT) population.
  years | 49.6 (10.88) | 51.9 (9.98) | 50.8 (10.48)
Age, Customized [Number; unit: Participants]
  < 30 years | 6 | 2 | 8
  Between 30 and 50 years | 44 | 44 | 88
  > 50 years | 64 | 68 | 132
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 33 | 60
  Male | 87 | 81 | 168

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response
Description: Clinical response defined as achieving all of the following 3 criteria on at least 2 consecutive visits or at the last on-treatment visit: Serum hepatitis B virus (HBV) DNA < 4 log10 copies/mL, normal Alanine transaminase (ALT) level (ALT ≤ Upper Limit of Normal (ULN)), and improvement (a 2- point or greater reduction in Child-Turcotte-Pugh (CTP) score) or stabilization (not more than a 1-point change in CTP score), compared to the baseline value. CTP scores range from 5-15, higher scores indicate more liver impairment. For Improvement/Stabilization, either of the individual criteria were met.
Time Frame: From Baseline to Week 52
Population: The analysis was on the intention-to-treat (ITT) population.
Measure: Number; unit: Participants
Arm/Group | Telbivudine 600 mg | Lamivudine 100 mg
Number analyzed (Participants) | 114 | 114
Participants
  Clinical Response | 65 | 62
  HBV DNA < 4log10copies/mL | 85 | 82
  Normal ALT | 78 | 81
  Improvement/stabilization in CTP | 96 | 96
  Improvement in CTP (reduction ≥ 2) | 34 | 43
  Stabilization in CTP (absolute change ≤ 1) | 56 | 48

2. Secondary Outcome: Time to Initial Clinical Response
Description: Time to Clinical Response defined as the number of days elapsed from the baseline visit to achieving initial Clinical Response.
Time Frame: From Baseline to Week 104
Population: The analysis was on intention-to-treat (ITT) population. Only the observed time to initial clinical response was summarized.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Telbivudine 600 mg | Lamivudine 100 mg
Number analyzed (Participants) | 95 | 92
Days | 137.5 (126.14) | 125.2 (111.24)

3. Secondary Outcome: Duration of Initial Clinical Response
Description: Kaplan-Meier method was used. The duration was calculated as: date of last visit before initial loss of clinical response - date of initial clinical response occurred+1. If a patient did not lose clinical response, it was then censored at the efficacy overall censoring date.
Time Frame: Baseline to Week 104
Population: The analysis was on intention-to-treat (ITT) population. Only patients who achieved clinical response were considered.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Telbivudine 600 mg | Lamivudine 100 mg
Number analyzed (Participants) | 95 | 92
Days | 473.1 (26.13) | 456.3 (24.97)

4. Secondary Outcome: Number of Participants With Improvement, Stabilization, and Worsening in Child-Turcotte-Pugh (CTP) Score at Week 52 and Week 104
Description: Child-Turcotte-Pugh (CTP) uses 2 clinical variables, ascites and encephalopathy, and 3 laboratory parameters, serum bilirubin, albumin, and prothrombin time. Each variable is assigned a score from 1 to 3, with the combined score comprising the CTP score range of 5 to 15 points. Higher scores indicate more impaired liver function. "Worsening" of CTP score was defined as a 2-point or greater increase from baseline, "improvement" in CTP score was defined as a 2-point or greater reduction from baseline, and "stabilization" of CTP score was defined as a change of 1-point or less from baseline.
Time Frame: From Baseline to weeks 52 and 104
Population: The analysis was done per intention-to-treat (ITT) population. Last Observation Carried Forward (LOCF) was utilized for missing data, with the exception of missing observations due to treatment failure, death or AE, which were imputed as "worsening" CTP.
Measure: Number; unit: Participants
Arm/Group | Telbivudine 600 mg | Lamivudine 100 mg
Number analyzed (Participants) | 114 | 114
Participants
  Improvement At Week 52 | 36 | 44
  Stabilization At Week 52 | 60 | 52
  Worsening At Week 52 | 18 | 18
  Improvement At Week 104 | 44 | 46
  Stabilization At Week 104 | 42 | 38
  Worsening At Week 104 | 28 | 30

5. Secondary Outcome: Number of Participants With Improvement, Stabilization, and Worsening in a Modified (3-component) CTP Score
Description: Modified CTP was calculated using the 3 biochemical-components (serum bilirubin, albumin, and prothrombin). Total scores range from 3-9; higher scores indicate more liver impairment. Improvement was defined as 2-point or greater reduction in score from baseline. Stabilization comprises a score change of 1-point or less from baseline. Worsening of CTP score was defined as a 2-point or greater increase from baseline. The rationale for assessing changes in this modified (3-component) CTP score is that this maneuver removed the two subjective components of CTP scoring (ascites and encephalopathy).
Time Frame: Baseline and Week 104
Population: The analysis was done on the intention-to-treat (ITT) population. Last Observation Carried Forward (LOCF) was utilized for missing data, with the exception of missing observations due to treatment failure, death or AE, which were imputed as "worsening" CTP.
Measure: Number; unit: Participants
Arm/Group | Telbivudine 600 mg | Lamivudine 100 mg
Number analyzed (Participants) | 114 | 114
Participants
  Improvement at Week 104 | 30 | 31
  Stabilization at Week 104 | 57 | 54
  Worsening at Week 104 | 27 | 29

ADVERSE EVENTS:
Description: Adverse event data is provided for the "on- treatment" period - i.e. any AEs started in the period of first dose date to last dose date + 30 days (all inclusive). For follow-up period, no individual preferred terms were reported in any treatment group. Hence, AE for follow-up period is not included here.
Arm/Group | Telbivudine 600 mg | Lamivudine 100 mg
Serious Adverse Events (participants affected / at risk) | 59/115 | 68/116
Other Adverse Events (participants affected / at risk) | 99/115 | 97/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telbivudine 600 mg (N=115) | Lamivudine 100 mg (N=116)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 11 | 2
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrage (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 3 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 7 | 3
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Death (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Hernia (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 1
Pitting oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Biloma (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 2
Hepatic dysplasia (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 2
Hepatorenal syndrome (Hepatobiliary disorders) | 3 | 1
Jaundice (Hepatobiliary disorders) | 1 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 2
Bacteraemia (Infections and infestations) | 1 | 1
Bronchitis acute (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 5 | 1
Dental caries (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 4
Hepatitis B (Infections and infestations) | 0 | 2
Necrostising fasciitis (Infections and infestations) | 0 | 1
Otitis media chronic (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 8 | 7
Pneumonia (Infections and infestations) | 1 | 3
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 8 | 0
Septic shock (Infections and infestations) | 3 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Subdiaphragmatic abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 3
Viral infection (Infections and infestations) | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Alpha 1 foetoprotein increased (Investigations) | 0 | 1
Ammonia increased (Investigations) | 1 | 0
Blood creatine phosphikinase increased (Investigations) | 0 | 1
Blood pressure systolic (Investigations) | 0 | 1
Transplant evaluation (Investigations) | 0 | 1
Viral load increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 12
Cerebellar infarction (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Coma hepatic (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 3 | 2
Hemiparesis (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 15 | 13
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Proststitis (Reproductive system and breast disorders) | 2 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Vaginal Prolapse (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemorrhoid operation (Surgical and medical procedures) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telbivudine 600 mg (N=115) | Lamivudine 100 mg (N=116)
Anaemia (Blood and lymphatic system disorders) | 6 | 7
Splenomegaly (Blood and lymphatic system disorders) | 6 | 7
Abdominal discomfort (Gastrointestinal disorders) | 3 | 10
Abdominal distension (Gastrointestinal disorders) | 23 | 14
Abdominal pain (Gastrointestinal disorders) | 12 | 14
Abdominal pain upper (Gastrointestinal disorders) | 6 | 10
Ascites (Gastrointestinal disorders) | 40 | 41
Constipation (Gastrointestinal disorders) | 9 | 9
Diarrhoea (Gastrointestinal disorders) | 15 | 16
Dyspepsia (Gastrointestinal disorders) | 15 | 12
Nausea (Gastrointestinal disorders) | 10 | 7
Varices Oesophageal (Gastrointestinal disorders) | 6 | 4
Vomiting (Gastrointestinal disorders) | 8 | 3
Asthenia (General disorders) | 5 | 12
Fatigue (General disorders) | 16 | 14
Oedema peripheral (General disorders) | 33 | 21
Pitting oedema (General disorders) | 13 | 12
Pyrexia (General disorders) | 20 | 17
Jaundice (Hepatobiliary disorders) | 15 | 11
Nasopharyngitis (Infections and infestations) | 5 | 9
Upper respiratory tract infection (Infections and infestations) | 17 | 12
Blood creatine phosphokinase increased (Investigations) | 7 | 2
Anorexia (Metabolism and nutrition disorders) | 6 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 8
Muscle cramp (Musculoskeletal and connective tissue disorders) | 6 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 5
Dizziness (Nervous system disorders) | 7 | 9
Encephalopathy (Nervous system disorders) | 6 | 6
Headache (Nervous system disorders) | 8 | 11
Hepatic Encephalopathy (Nervous system disorders) | 7 | 7
Insomnia (Psychiatric disorders) | 11 | 9
Gynaecomastia (Reproductive system and breast disorders) | 16 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 12
Spider Naevus (Skin and subcutaneous tissue disorders) | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.